CLINICAL TRIAL: NCT01472575
Title: An Observational, Cross-sectional, Cohort Study to Assess the Impact of the Rotavirus Vaccine Introduction on Severe Gastroenteritis in South Australian Children
Brief Title: Impact of Rotavirus Vaccine Introduction for South Australian Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Associate Professor Helen Marshall (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Associate Professor Helen Marshall, Director, Vaccinology and Immunology Research Trials Unit, Women's and Children's Hospital, Australia
Organization: Women's and Children's Hospital, Australia (Other Government)
Other Study IDs: 38070; 38070 (Other Grant/Funding Number: IISP 38070 Merck)
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Viral Gastroenteritis Due to Rotavirus; Gastroenteritis
Keywords: rotavirus; gastroenteritis; vaccination; hospitalisation
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre- rotavirus vaccination introduction: Children aged 0-less than 6 years of age admitted to hospital in South Australia with ICD10-AM separation codes consistent with rotaviral infection or gastroenteritis of any cause during the period 01May2005-30Apr2007 (pre vaccine introduction)
- post rotavirus vaccine introduction: Children aged 0-less than 6 years of age admitted to hospital in South Australia with ICD10-AM separation codes consistent with rotaviral infection or gastroenteritis of any cause during the period 01May2009-30Apr2011 (post vaccine introduction)

SUMMARY:
This project aims to assess the impact of rotavirus vaccine introduction on severe gastroenteritis in South Australian children. Prevalence of rotavirus coded hospitalisations and all-cause gastroenteritis hospitalisations will be compared for a two year period prior to introduction of the vaccine and a two year period following introduction of the vaccine. Severity of rotavirus coded admissions during the periods will also be assessed.

Hypotheses:

1. Introduction of the rotavirus vaccine will result in an 80% reduction in hospitalisations for rotavirus positive gastroenteritis (ICD code A0.80) in children less than two years of age.
2. Introduction of rotavirus vaccine will result in an 80% reduction in Paediatric Emergency presentations for rotavirus positive gastroenteritis in children under two years of age.
3. Introduction of the rotavirus vaccine will result in a 50% reduction in hospitalisations for all cause gastroenteritis (ICD codes A0.00-A0.90) in children less than two years of age.
4. Introduction of the rotavirus vaccine will result in a 50% reduction in Paediatric Emergency presentations for all cause gastroenteritis in children less than two years of age.
5. Introduction of rotavirus vaccine will result in a reduction in hospitalisation and Paediatric Emergency presentations in children aged four and five years with rotavirus positive gastroenteritis (unvaccinated cohort).
6. There will be no difference in severity of disease as scored by the Vesikari and/or clark severity score prior to and post introduction of rotavirus vaccine

DETAILED DESCRIPTION:
This project aims to assess vaccine effectiveness in the field following introduction of the rotavirus vaccine in South Australian children. It is important to confirm the benefits of the vaccine post licensure to ensure the best health care options for children. Between July 2007 - June 2008 at the Women's and Children's Hospital, there were approximately 2000 gastroenteritis patient samples analysed, with approximately 200 of these confirmed as rotavirus positive (10%). The current vaccines available in Australia (Rotarix® and RotaTeq® ) are licensed for administration in infants up to six months of age as safety data is not yet available for older children. It is therefore important to determine whether vaccination according to the current Australian Standard Vaccination Schedule can also demonstrate a positive change (less disease and less severe disease) in the burden of rotavirus disease in older unvaccinated children.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 0-less than 6 years of age admitted to SA hospital with ICD10-AM separation codes consistent with rotaviral infection or gastroenteritis of any cause.
* for severity component, only admissions to the Women's and Children's Hospital will be examined

Exclusion Criteria:

* nosocomial rotaviral infections (defined as onset >48 hours post admission date) will be reported separately in the severity analysis

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: males and females aged 0-less than 6 years of age admitted to SA hospital with ICD10-AM separation codes consistent with rotaviral infection or gastroenteritis of any cause.
  - for severity component, admissions to the Women's and Children's Hospital will be examined.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in prevalence of rotavirus coded hospital admissions before and after introduction of rotavirus vaccination | 2 years prior to vaccine introduction (01May2005-30Apr2007) and 2 years post vaccine introduction (01May2009-30Apr2011)

SECONDARY OUTCOMES:
Change in prevalence of all-cause gastroenteritis coded hospital admissions before and after rotavirus vaccination introduction | 2 years prior to vaccine introduction (01May2005-30Apr2007) and 2 years post vaccine introduction (01May2009-30Apr2011)
Change in proportion of admissions scored as severe (scored by severity index) for rotavirus coded hospital admissions before and after introduction of rotavirus vaccination | 2 years prior to vaccine introduction (01May2005-30Apr2007) and 2 years post vaccine introduction (01May2009-30Apr2011)

CONTACTS AND LOCATIONS:
Overall Officials: Helen S Marshall, MBBS MD MPH, Principal Investigator — Women's and Children's Health Network
Locations (1):
- Women's and Children's Hospital, North Adelaide, South Australia, Australia

REFERENCES:
- [Result] Clarke MF, Davidson GP, Gold MS, Marshall HS. Direct and indirect impact on rotavirus positive and all-cause gastroenteritis hospitalisations in South Australian children following the introduction of rotavirus vaccination. Vaccine. 2011 Jun 24;29(29-30):4663-7. doi: 10.1016/j.vaccine.2011.04.109. Epub 2011 May 14. PMID 21575665